CLINICAL TRIAL: NCT01473355
Title: An Open, Prospective, Multi-center Study to Evaluate OsseoSpeed™ TX Single Implant 3 mm Diameter in the Anterior Mandible. A 3-years Follow-up Study.
Brief Title: Study on OsseoSpeed™ TX Narrow Implants in the Lower Jaw in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-0003
Record Dates: First submitted 2011-11-15; First posted 2011-11-17 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Partially Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous, Partially

ARMS (1):
- OsseoSpeed™ TX (Experimental): OsseoSpeed™ TX narrow implants (diameter 3 mm) in lengths of 11-15 mm
  Interventions: Device: OsseoSpeed™ TX

INTERVENTIONS:
Device: OsseoSpeed™ TX — OsseoSpeed™ TX narrow implants (diameter 3 mm) of lengths 11-15 mm

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of OsseoSpeed™ TX 3mm diameter implant in a Chinese population by evaluation of marginal bone level alteration, implant stability and implant survival in the posterior mandible up to 3 years after loading. Hypothesis: Early loading of the 3 mm implant is a safe and predictable procedure.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent
2. Aged 20-75 years at enrolment
3. History of edentulism in the study area of at least two months
4. Presence of natural teeth, partial prosthesis and/or implants in the opposite jaw in contact with the planned crowns
5. Deemed by the investigator to have a bone height and width suitable for 3.0 mm diameter study implant
6. Deemed by the investigator as likely to present an initially stable implant situation

Exclusion Criteria:

1. Unlikely to be able to comply with study procedures, as judged by the investigator
2. Uncontrolled pathologic processes in the oral cavity
3. Known or suspected current malignancy
4. History of radiation therapy in the head and neck region
5. History of chemotherapy within 5 years prior to surgery
6. Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration, as deemed by the investigator
7. Uncontrolled diabetes mellitus
8. Corticosteroids or any other medication that could influence post-operative healing and/or osseointegration
9. Smoking more than 10 cigarettes per day
10. Present alcohol and/or drug abuse
11. Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
12. Previous enrollment in the present study
13. Simultaneous participation in another clinical study, or participation in a clinical study during the last weeks prior to enrollment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping Gong, Prof, Principal Investigator — Sichuan University
Locations (3):
- China (3):
  - School of Stomatology, JiLin University, Hospital of Stomatology, Changchun
  - Sichuan University, Chengdu
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Groups:
- OsseoSpeed™ TX: OsseoSpeed™ TX narrow implant (diameter 3 mm) in lengths of 11-15 mm
Period: Overall Study
Arm/Group | OsseoSpeed™ TX
Started | 45; 75 Implants
Completed | 39; 65 Implants
Not Completed | 6; 10 Implants
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 45
Number analyzed (Implants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 33
Region of Enrollment [Number; unit: participants]
  China | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Survived Implants
Description: Implant survival rate evaluated by clinically and radiographically counting the number of implants remaining in function
Time Frame: Measured at the 3 year follow-up after implant loading.
Population: All participants treated with at least one study implant.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 45
Number analyzed (Implants) | 75
Implants | 74

2. Secondary Outcome: Marginal Bone Level Alteration
Description: Marginal bone level determined from radiographs and expressed as the distance from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal bone level expressed in millimeters at the 3 year follow-up visit compared to values obtained at delivery of permanent restoration i.e. loading (baseline).
Time Frame: Measured at the 3 year follow-up after implant loading.
Population: 39 subjects (65 implants) completed the 3-year follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 34 subjects (60 implants). Three of the radiographs were not possible to evaluate, giving an overall number of 32 subjects (57 implants) as basis for the Marginal Bone Level analysis.
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 32
Number analyzed (Implants) | 57
millimeter | -0.02 (0.80)

3. Secondary Outcome: Number of Stable Implants
Description: Implant stability evaluated clinically/manually (recorded as stable yes/no).
Time Frame: Measured at the 3 year follow-up after implant loading.
Population: 39 subjects (65 implants) completed the 3-year follow-up visit. Analysis of implant stability was performed on the all patients treated population.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 39
Number analyzed (Implants) | 65
Implants | 65

4. Secondary Outcome: Evaluation of the Periimplant Mucosa Condition - By Assessment of PPD
Description: Condition of the periimplant mucosa by assessment of probing pocket depth (PPD).
  Change in pocket depth expressed in millimeters at the 3-year follow-up visit, compared to values obtained at delivery of permanent restoration, i.e. loading (baseline).
  Negative value = increased pocket depth.
Time Frame: Measured at the 3 year follow-up after implant loading.
Population: 39 subjects (65 implants) completed the 3-year follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 34 subjects (60 implants) for the PPD analysis.
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 34
Number analyzed (Implants) | 60
millimeter | -0.03 (0.59)

5. Secondary Outcome: Evaluation of the Periimplant Mucosa Condition - By Assessment of BoP
Description: Condition of the periimplant mucosa by assessment of Bleeding on Probing (BoP). Presented as % of implants that show presence of bleeding on probing at time of the 3-year follow-up visit.
Time Frame: Measured at the 3 year follow-up after implant loading.
Population: 39 subjects (65 implants) completed the 3-year follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 34 subjects (60 implants) for the BoP analysis.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 34
Number analyzed (Implants) | 60
Implants | 33

6. Secondary Outcome: Presence of Plaque
Description: Occurence of plaque around the study implant. Presented as number of implants that show presence of plaque at time of the 3 years follow-up visit after implant loading.
Time Frame: Measured at the 3 year follow-up after implant loading.
Population: 39 subjects (65 implants) completed the 3-year follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 34 subjects (60 implants) for the plaque analysis.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 34
Number analyzed (Implants) | 60
Implants | 49

ADVERSE EVENTS:
Time Frame: 3 year
Arm/Group | OsseoSpeed™ TX
Serious Adverse Events (participants affected / at risk) | 2/45
Other Adverse Events (participants affected / at risk) | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed™ TX (N=45)
Fracture left leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Possible ablepsia of right eye (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less